CLINICAL TRIAL: NCT06919731
Title: PLATELET-ASSOCIATED TISSUE FACTOR AS A NEW BIOMARKER FOR THROMBOTIC RISK STRATIFICATION IN PATIENTS WITH CORONARY ARTERY DISEASE.
Brief Title: PLATELET TISSUE FACTOR AS BIOMARKER OF THROMBOTIC RISK IN CORONARY ARTERY DISEASE PATIENTS (TRIT-ONE)
Acronym: TRIT-ONE
Status: Completed | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: R1436/21-CCM 1508
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases
Keywords: Platelet; Tissue Factor; Biomarker; coronary artery diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: whole blood flow cytometry analisys — Evaluation of platelet prothrombotic potential through a flow-cytometry analysis of platelet activation marker expression, including P-selectin, aGPIIbIIIa and TF, as well as platelet-leukocyte aggregate formation.

SUMMARY:
Enhancing thrombotic risk stratification in patients with coronary artery disease (CAD) is crucial for the prevention and management of cardiovascular disease. Existing risk scores, which predict mortality risk and/or the likelihood of adverse cardiovascular events, are based on clinical and laboratory parameters. However, none of these scores incorporates the elevated platelet activation observed in CAD, a critical factor influencing disease progression.

Over the past two decades, research has consistently shown that activated platelets play a pivotal role in plaque formation. These platelets, together with fibrin, form the primary components of thrombi that obstruct coronary arteries, making them central to the pathogenesis of coronary syndromes. Published studies have highlighted how platelet activation triggers the expression of Tissue Factor (TF), a key glycoprotein involved in blood coagulation and thrombotic complications in atherosclerosis. Notably, in patients with coronary syndrome, platelet TF expression is significantly higher than in healthy individuals. The functional ability of platelet TF to generate thrombin further enhances the pro-thrombotic potential of these platelets, underscoring their critical role in thrombus formation.

The objective of this study is to validate the predictive value of platelet Tissue Factor (TF) for cardiovascular events in a cohort of secondary prevention patients treated with antiplatelet drugs, including clopidogrel, ticagrelor, prasugrel, and/or aspirin. The primary endpoint is the assessment of all-cause mortality and cardiovascular death, over a 5-year follow-up period from admission.

ELIGIBILITY:
Inclusion Criteria:

patients of either sex, aged 18 years or older, with a diagnosis of acute or stable coronary syndrome, treated with anti-platelet drugs (aspirin and/or clopidogrel, prasugrel and ticagrelor) as per guidelines

Exclusion Criteria:

pregnant subjects (self-declared); subjects who have received blood transfusions in the last 30 days; subjects over 89 years of age; subjects with hereditary platelet disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited among patients admitted to the Cardiology Units of the Centro Cardiologico Monzino IRCCS
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality and cardiovascular death | From enrollment to the end of 5-follow-up
  Assessment of all-cause mortality and cardiovascular death over a 5-year follow-up period from enrollment.